CLINICAL TRIAL: NCT02894333
Title: The Process of Sensory Anticipation in Patients With PARKINSON's Disease
Brief Title: Action-effect Anticipation in Patients With Parkinson's Disease : A Study of the Sensory Attenuation Marker.
Acronym: IDEOMOT
Status: Terminated | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JBL_2014-30
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Action-effect prediction; Sensory attenuation; Voluntary action
MeSH Terms: conditions — Parkinson Disease | interventions — Behavior Observation Techniques

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Patients with Parkinson's disease
  Interventions: Behavioral: behavioral observation

INTERVENTIONS:
Behavioral: behavioral observation

SUMMARY:
The ideomotor theory of action control is considered to be central to the understanding of human voluntary action. According to the ideomotor theory, an action is represented in terms of its desired sensory effects and actions are selected by internally activating these effect representations. Recent imagery and behavioral studies showed that this anticipated representation of action-effects triggered a "sensory attenuation", meaning a decrease of perceptive performances or a decrease of sensory event-related potentials (ERP) for an expected event. Thus, the sensory attenuation constitutes a relevant behavioral tool to investigate sensory anticipation impairment in patients with Parkinson's disease. In a behavioral paradigm, patients and matched control participants have to perform a perceptive task on predicted visual action-effects mixed with mispredicted visual action effects. Performances should be better in mispredicted visual action effects for control participants only.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Normal or corrected vision

Exclusion Criteria:

* Other pathology or neurological or psychiatric history
* Known pregnancy or breastfeeding
* Absence of affiliation to the French Social Security
* Person under legal protection
* Patient's opposition to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
median score | baseline
  scores measured with the Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Fondation Adolphe de Rothschild, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris